CLINICAL TRIAL: NCT06212050
Title: Investigator Initiated Multicenter Study to Evaluate the Feasibility, Safety and Effectiveness of the ACURATE neo2 Transcatheter Heart Valve for Severe Bicuspid Aortic Stenosis - The Neo2 BAV Registry
Brief Title: Feasibility, Safety, and Effectiveness of the ACURATE neo2 Transcatheter Heart Valve for Severe Bicuspid Aortic Stenosis
Acronym: Neo2BAV
Status: Enrolling by invitation | Type: Observational
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Galway University Hospitals (Unknown); CORRIB Research Centre for Advanced Imaging and Core Lab, Galway, Ireland (Unknown); Karolinska University Hospital (Other); Kerckhoff Heart Center (Other)
Responsible Party: Principal Investigator, Professor Osama SOLIMAN, Professor of Cardiovascular Research, National University of Ireland, Galway, Ireland
Other Study IDs: C.A. 2961
Record Dates: First submitted 2023-11-08; First posted 2024-01-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Aortic Stenosis; Transcatheter Aortic Valve Implantation; Bicuspid Aortic Valve; Transcatheter Aortic Valve Replacement
Keywords: ACURATE neo2; Aortic stenosis; Bicuspid Aortic valve
MeSH Terms: conditions — Aortic Valve Stenosis; Bicuspid Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe symptomatic BAV stenosis: Patients with severe symptomatic BAV stenosis who underwent TAVI using the ACURATE neo2 THV.
  Interventions: Device: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — TAVI in patients with severe BAV stenosis using ACURATE neo2
  Other Names: ACURATE neo2 Aortic valve system

SUMMARY:
The goal of the NEO2 BAV registry is to investigate the safety, effectiveness, and clinical performance of TAVI using the ACURATE neo2 valve in patients with severe BAV stenosis.

The clinical, procedural, and imaging characteristics will be collected from patients with severe BAV stenosis, regardless of the phenotype, and treated with TAVI using the ACURATE neo2 bioprosthesis worldwide.

DETAILED DESCRIPTION:
As the use of TAVI in BAV anatomy expands, it is important to systematically evaluate clinical outcomes from various THV technologies among BAV patients. It is essential to consider short-, and longer-term events among patients with BAV undergoing TAVI. Short-term outcomes of interest include THV embolization, PVL, residual transvalvular gradients and patient prosthesis mismatch, aortic root rupture, the requirement for new PPI, and stroke. Longer-term term clinical events of interest include quality of life, THV durability, freedom from reintervention, maintained coronary access, the possibility of redo-TAVI, and mortality.

The ACURATE neo2 THV has design features that make it possible to successfully treat severe BAV stenosis and yield optimal short- and longer-term outcomes. A new active sealing skirt is designed to minimize residual PVL; this is especially relevant given the presence of severe calcifications in BAV. The supra-annular leaflet position is also likely to provide excellent haemodynamics and durability since they sit above the heavily calcified native valve leaflet calcification. The upper crown and stabilizing arches and the top-down deployment of the ACURATE neo2 should reduce the risk of device embolization. It is unclear however if the self-expanding frame of the neo2 has the optimal radial force to treat patients with severe calcification.

The plan is to collect systematic clinical, procedural, and imaging data on a large series of patients with severe symptomatic BAV stenosis who underwent TAVI using the ACURATE neo2 THV. This information will show if the ACURATE neo2 is suitable to treat BAV morphology and determine if there are specific BAV subtypes that are more suitable for alternative treatment strategies. It is also envisaged that this study will inform the procedural execution of ACURATE neo2 THV in BAV morphology and inform future iteration design of the ACURATE neo THV series.

All imaging data (Echocardiography, angiography, aortography and MSCT) will be meticulously analyzed in an independent imaging Core Lab (CORRIB Core Lab, University of Galway, Galway, Ireland).

The in-depth imaging analysis will allow the identification of patients that are suitable for TAVI using the ACURATE neo2 system and highlight patient or procedural features that render TAVI at elevated risk of adverse outcomes. Furthermore, a mechanistic understanding of the device-host interaction will be examined on post-TAVI multislice computed tomography (MSCT) and other available post-TAVI imaging studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with severe AS and any BAV phenotype and indicated for TAVI based on the local heart team decision.
* Patient treated with ACURATE neo2 THV.

Exclusion Criteria:

* Failure to obtain the patient's consent
* Failure to obtain the follow-up clinical data or cardiac imaging required for the study primary endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe BAV stenosis and treated with TAVI using ACURATE neo2 THV.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
VARC-3 device success | 30-Day
  1. Number of patients with technical success.
  2. Number of patients with death from any cause.
  3. Number of patients with surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication.
  4. Number of patients with intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate AR), defined as the presence of all of the following:
VARC-3 early safety | 30-Day
  1. Number of patients with death from any cause.
  2. Number of patients with stroke.
  3. Number of patients with VARC type 2-4 bleeding.
  4. Number of patients with major vascular, access-related, or cardiac structural complication.
  5. Number of patients with acute kidney injury stage 3 or 4.
  6. Number of patients with moderate or severe aortic regurgitation
  7. Number of patients with new pacemaker due to procedure related conduction abnormalities
  8. Number of patients with surgery or intervention related to the device

SECONDARY OUTCOMES:
VARC-3 clinical efficacy (at 1 year and thereafter) | 1-year
  1. Number of patients with death from any cause.
  2. Number of patients with stroke.
  3. Number of patients with hospitalization (procedure or Valve related causes).
Valve-related long-term clinical efficacy (at 5 years and thereafter) | 5-year
  1. Number of patients with bioprosthetic Valve Failure (defined as: Valve related mortality OR Aortic valve re-operation/re-intervention or Stage 3 hemodynamic valve deterioration)
  2. Number of patients with stroke.
  3. Number of patients with VARC Type 2-4 bleeding secondary to or exacerbated by antiplatelet or anticoagulant agents, used specifically for valve-related concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Mylotte, MD, PhD, Principal Investigator — University of Galway, Galway University Hospital; Andreas Ruck, MD, Principal Investigator — Karolinska University Hospital; Won-Keun Kim, MD, Principal Investigator — Kerckhoff Heart and Lung Centre; Osama Soliman, MD, PhD, Principal Investigator — University of Galway, Galway University Hospital
Locations (3):
- Kerckhoff Heart and Lung Centre, Bad Nauheim, Germany
- Galway University Hospital, Galway, Ireland
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet